CLINICAL TRIAL: NCT03476447
Title: Rescuing the Microbiome Effectively With Different Doses of B. Infantis in Infants (The REMEDI Study)
Brief Title: Rescuing the Microbiome Effectively With Different Doses of B. Infantis in Infants
Acronym: REMEDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evolve BioSystems, Inc. (Industry)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1166403
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Gut Microbiome
MeSH Terms: interventions — Lactose

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled and randomized 1:1:1:1 to the following treatment arms (daily dose of B. infantis EVC001): high dose, medium dose, low dose, and placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators and data evaluators will be blinded to the treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High dose B. infantis EVC001 (Active Comparator): 10 participants will receive powdered B. infantis EVC001 at a high dose per daily oral feeding
  Interventions: Other: B. infantis EVC001
- Medium dose B. infantis EVC001 (Active Comparator): 10 participants will receive powdered B. infantis EVC001 at a medium dose per daily oral feeding
  Interventions: Other: B. infantis EVC001
- Low dose B. infantis EVC001 (Active Comparator): 10 participants will receive powdered B. infantis EVC001 at a low dose per daily oral feeding
  Interventions: Other: B. infantis EVC001
- Lactose Placebo (Placebo Comparator): 10 participants will receive powdered lactose per daily oral feeding
  Interventions: Other: Lactose

INTERVENTIONS:
Other: B. infantis EVC001 — A once-daily oral feeding of B. infantis EVC001 will be mixed with breast milk and provided to infants for 28 consecutive days.
  Arms: High dose B. infantis EVC001; Low dose B. infantis EVC001; Medium dose B. infantis EVC001
Other: Lactose — A once-daily oral feeding of a lactose placebo will be mixed with breast milk and provided to infants for 28 consecutive days.
  Arms: Lactose Placebo

SUMMARY:
The REMEDI Study is a single-center, prospective, double-blind, randomized, placebo-controlled trial of multiple doses of B. infantis EVC001 supplementation in healthy term breastfed infants.

DETAILED DESCRIPTION:
Mother-infant dyads will be enrolled when the infant is 2-4 months of age. A 1-week lead-in period will be utilized to collect baseline microbiome samples and for the completion of daily and weekly feeding and health logs. Subjects that meet eligibility criteria on Day 7 will be randomized into 1 of 4 treatment arms. Supplementation will begin on Day 8 and will continue for a total of 28 consecutive days. Subjects will be followed for an additional 4 weeks after the cessation of the supplement. The total duration of the study will be approximately 9 weeks. Infant stool and urine samples, as well as maternal breast milk samples, will be collected on multiple occasions during the study. Mothers will be asked to complete questionnaires and health logs during the course of the study as well.

ELIGIBILITY:
Inclusion Criteria:

* Age of subjects: Infants: 60 to 125 days old, Mothers: 21 years old and greater
* Mother-infant dyads who live within a 40-mile radius from the clinical site
* Infants predominately breastfed with maternal intent to continue exclusive breastfeeding for at least 9 additional weeks
* Term infants born >37 weeks gestation
* Healthy infants without medical complications
* Generally healthy women
* Mothers who are willing to refrain from feeding their infants infant formula, solid foods, and probiotic or iron supplements (confounding variables of the intestinal microbiome) before the end of the study

Exclusion Criteria:

* Mothers diagnosed with any metabolic, endocrine, liver, or kidney disease, any autoimmune disease, cirrhosis, hepatitis C, HIV, AIDs, cancer, obesity (pre-pregnancy BMI >34.9 kg/m2), Crohn's disease, heart disease, type 1 or type 2 diabetes (type 1 diabetes is acceptable if mother's blood glucose has been well-regulated)
* Infants born in a multiple birth
* Infants born with medical complications such as: respiratory distress syndrome or birth defects
* Infants with any GI tract abnormalities
* Infants who have taken antibiotics within 4 weeks of enrollment or during the Lead-in Period
* Infants who have taken iron supplements within 4 weeks of enrollment or during the Lead-in Period
* Infants who have consumed any infant formula within 4 weeks of enrollment or more than 10 times between birth and enrollment or during the Lead-in Period
* Infants whose parents plan to feed them any infant formula any time throughout the duration of the study
* Infants who have consumed any probiotics containing B. infantis since birth
* Infants who have consumed any Bifidobacterium-containing probiotics within 4 weeks of enrollment or during the Lead-in Period
* Infants whose parents plan to administer probiotics to them any time throughout the duration of the study (not including the study supplement)
* Infants who have consumed any solid foods or beverages between birth and enrollment or during the Lead-in Period (liquid medicines, supplements, and sugar water are ok)
* Infants whose parents plan to feed them solid foods or beverages any time throughout the duration of the study
* Infants whose mothers have changed their minds about their plans to exclusively breastfeed for at least 8 additional weeks by Day 7
* For infants born vaginally, maternal intake of probiotics containing B. infantis during the last trimester of pregnancy
* Mother-infant dyads who live in more than one location
* Infants who have been diagnosed with any medical or nutritional condition that would require iron supplementation
* Mothers who smoked cigarettes during pregnancy, currently smoke, or plan to initiate smoking during the study duration
* Anyone the investigator feels isn't an applicable subject

Ages: 2 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Fecal B. infantis levels in infants at 28 days - difference between B. infantis and placebo | 28 days
  The difference in levels of infant fecal B. infantis (as measured by B. infantis qPCR) between B. infantis EVC001 supplementation and placebo supplementation on Day 28.

SECONDARY OUTCOMES:
Fecal B. infantis levels in infants at 28 days - difference between B. infantis doses | 28 days
  The differences between B. infantis EVC001 doses on levels of infant fecal B. infantis (as measured by B. infantis qPCR) on Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Smilowitz, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Brien CE, Frese SA, Cernioglo K, Damian-Medina K, Mitchell RD, Casaburi G, Melnyk RA, Henrick BM, Smilowitz JT. Randomized, placebo-controlled trial reveals the impact of dose and timing of Bifidobacterium infantis probiotic supplementation on breastfed infants' gut microbiome. mSphere. 2025 Dec 22:e0051825. doi: 10.1128/msphere.00518-25. Online ahead of print. PMID 41427732